CLINICAL TRIAL: NCT02096406
Title: COMParison of Angiotensin Converting Enzyme Inhibitor managemenT Strategies Prior to Coronary Artery Bypass Surgery (the COMPACT Trial): a Pilot Randomized Controlled Registry Study
Brief Title: Outcomes of Angiotensin Converting Enzyme Inhibitor Management Strategies Prior to Coronary Artery Bypass
Acronym: COMPACT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Principal Investigator, Sean van Diepen, Assistant Professor of Critical Care Medicine and Cardiology, University of Alberta
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00042749
Record Dates: First submitted 2014-03-17; First posted 2014-03-26 (Estimated); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: Coronary Artery Disease
Keywords: Coronary artery disease; Coronary artery bypass grafting; angiotensin converting enzyme inhibitor; angiotensin receptor blocker; Surgical valve repair; Valve Replacement
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ACE/ARB Continuation (Other): ACE/ARB will be continued up to and including the morning of surgery.
  Interventions: Drug: ACE/ARB continuation
- ACE/ARB withdrawal (Other): ACE/ARB will be discontinued medication 48 hours prior to surgery
  Interventions: Drug: ACE/ARB withdrawal

INTERVENTIONS:
Drug: ACE/ARB continuation — ACE/ARB will be taken the morning of surgery with a sip of water
  Arms: ACE/ARB Continuation
Drug: ACE/ARB withdrawal — ACE/ARB will be stopped 48 hours prior to surgery
  Arms: ACE/ARB withdrawal

SUMMARY:
Coronary artery disease is a leading cause of death, hospitalization, and health care costs in developed nations. Coronary revascularization with coronary artery bypass graft (CABG) surgery improves the long term survival in patients with diabetes and multi-vessel disease. Angiotensin converting enzyme inhibitors (ACE) and angiotensin receptor blockers (ARB) reduce mortality and subsequent cardiac events in patients with coronary artery disease undergoing CABG surgery when initiated at least 4 weeks pre-operatively. Observational data have suggested that pre-operative ACE administration is associated with an increased risk of post-operative vasoplegic shock, acute kidney injury, and mortality; however, other studies have failed to confirm these findings and further suggested ACE are associated with a reduced risk of peri-operative myocardial infarction. A single trial of 40 CABG patients randomized to pre-operative ACE withdrawal or continuation reported that the withdrawal group required significantly fewer vasopressors during cardiopulmonary bypass but more intravenous vasodilators post-operatively to control hypertension. Hence, it remains unclear whether ACEs should be held or continued immediately prior to CABG surgery and a survey of cardiac surgeons suggests that current clinical practice is divided. This pilot study aims to establish the feasibility of the study design and to determine the frequency of clinical endpoints among patients who continue and discontinue ACE prior to cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective or urgent isolated CABG and/or valvular repari or replacement surgery
* On an ACE or ARB for a minimum of 7 days

Exclusion Criteria:

* Emergency surgery
* Pre-operative shock (defined as systolic blood pressure < 90 mmHg, the need for any vasopressor or inotropic support, or a mechanical cardiac support device)
* Severe uncontrolled pre-operative hypertension (defined as blood pressure ≥ 200 mmHg systolic or ≥120mmHg diastolic mmHG or the pre-operative need for intravenous anti-hypertensive agents)
* ACE or ARB therapy < 7 days
* Any mineralocorticoid receptor antagonist therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2014-04; Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Adherence to the study protocol | From randomization to surgery
  Proportion of patients who adhere to ACE/ARB continuation or withdrawal as randomized
Feasibility of study enrollment | 30 dasys
  >50% of eligible patients are successfully enrolled in the trial
Feasibility of Study | 60 days
  >=95% completeness of outcomes

SECONDARY OUTCOMES:
Feasibility of the Study | 30 days
  Reasons for non-recruitment
Incidence of post operative Shock | 3 hours
  Post-operative shock (use of any intravenous vasopressors (norepinephrine, epinephrine, vasopressin, dopamine, and/or methylene blue) and mechanical support devices (left ventricular assist devices, intra-aortic balloon pumps, or extracorporeal membrane oxygenation) initiated within the first 3 hours of CVICU admission)
Duration of Shock | 7 days
  Post-operative shock (use of any intravenous vasopressors (norepinephrine, epinephrine, vasopressin, dopamine, and/or methylene blue) and mechanical support devices (left ventricular assist devices, intra-aortic balloon pumps, or extracorporeal membrane oxygenation) initiated within the first 3 hours of CVICU admission)
Vasopressors use | 7 days
  Number and maximum dose of vasopressors
Post operative intravenous anti-hypertensive use | 7 days
  The post-operative use intravenous vasodilators (nitroglycerine or nitroprusside)
Duration of intravenous vasodilator use | 7 days
  The post-operative duration intravenous vasodilators (nitroglycerine or nitroprusside)
Vasodilator use | 7 days
  The number and maximum dose of vasodilators
Incidence of vasoplegic shock | 4 hours
  Vasopressor administration for at lead 4 hours despite intravenous fluid administration
Pre-operative heart failure deterioration | 48 hours
  Any increase in diuretic dose in 48 hours prior to surgery
Post-operative acute kidney injury | 7 days
  Acute kidney injury defined as a doubling of serum creatinine within 7 days of surgery
Change in renal function | 7 days
  Difference between baseline and peak post-operative creatinine
Initiation of renal replacement therapy | 7 days
Peak post-operative troponin | 72 hours
  Peak post-operative troponin within 72 hours of surgery
Stroke | 30 days
  Incidence of any stroke within 30 days of surgery
In hospital Mortality | Participants will be followed for the duration of hospital stay, an expected average of 7 days

OTHER OUTCOMES:
ACE or ARB use at hospital discharge | Participants will be followed for the duration of hospital stay, an expected average of 7 days
Duration of post-operative mechanical ventilation | 7 days
  Time to extubation after admission to ICU
Cardiovascular ICU length of stay | Participants will be followed for the duration of the ICU stay, an expected average of 2 days
ICU readmission | Participants will be followed for the duration of hospital stay, an expected average of 7 days
  Incidence and cause of any ICU readmission after discharge to lower acuity ward post-operatively.

CONTACTS AND LOCATIONS:
Overall Officials: Sean van Diepen, MD, Msc, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta Hospital, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] van Diepen S, Norris CM, Zheng Y, Nagendran J, Graham MM, Gaete Ortega D, Townsend DR, Ezekowitz JA, Bagshaw SM. Comparison of Angiotensin-Converting Enzyme Inhibitor and Angiotensin Receptor Blocker Management Strategies Before Cardiac Surgery: A Pilot Randomized Controlled Registry Trial. J Am Heart Assoc. 2018 Oct 16;7(20):e009917. doi: 10.1161/JAHA.118.009917. PMID 30371293